CLINICAL TRIAL: NCT05692375
Title: Impact of the Save the Shame! Game on Advanced Life Support Knowledge of Nurses and Physicians in Intensive Care Medicine Settings, a Pilot Randomized Study
Brief Title: Impact of the Save the Shame! Game on Advanced Life Support Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E. (Other Government)
Collaborators: University of Minho (Other)
Responsible Party: Principal Investigator, Sara Santos Ribeiro, Principle investigator, Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 01
Record Dates: First submitted 2023-01-10; First posted 2023-01-20 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Intensive Care
Keywords: healthcare; gamification; education; advanced life support

STUDY DESIGN:
Intervention Model Description: The investigators developed an experimental approach, where we ensured randomization in sample identification and where a control group was present, favoring a strongest level of contribution to the evidence. This is a cross-sectional study with quantitative data collection following a Randomized Controlled Trial (RCT) design.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will be inveted to use the game. Two weeks were defined as the time to use the game. The use of the game can be seen by the coded digital record on its digital platform .
  Interventions: Other: Invitation to play the game "Save the shame!"
- Control (No Intervention): The control group neither used nor had access to the game.

INTERVENTIONS:
Other: Invitation to play the game "Save the shame!" — The experimental group was asked to use the game. Two weeks were defined as the time to use the game. The use of the game can be seen by the coded digital record on its digital platform . The control group neither used nor had access to the game. Afterwards both groups performed the ALS knowledge assessment test. It is a test with 20 multiple choice questions each scored as right (0.5 points) or wrong (0 points).
  Arms: Experimental

SUMMARY:
Gamification, listed by the European Resuscitation Council (ERC) as a learning process in its 2021 guidelines, is a new digital innovation tool that brings added value towards motivation that seems to reuse time in a creative way. The aim of this study is to evaluate the impact of the game "Save the shame!" on advanced life support (ALS) knowledge of nurses and physicians in intensive care medicine settings. This is a cross-sectional study following a mixed methodology. In its preliminary phase it follows a qualitative and exploratory methodology, with application of the E-Delphi technique for creation and validation of the "Save the shame! game and validation of the ALS knowledge test. The study subsequently follows the experimental methodology. The investigators expect to confirm the hypothesis that the game "Save the Shame!" has a positive impact on the skills training of health professionals in intensive care medicine settings in a Portuguese hospital center.

DETAILED DESCRIPTION:
Study Design The investigators developed an experimental approach, where randomization in sample identification was ensured and where a control group was present, favoring a strongest level of contribution to the evidence. This is a cross-sectional study with quantitative data collection following a Randomized Controlled Trial (RCT) design.

In order to carry out the proposed experimental study, it was necessary to create two essential elements in this process: the "Save the Same!" game and the ALS knowledge assessment test, which constitutes a data collection instrument necessary to test the research hypotheses.

Arms, Groups, and Interventions The population was defined as nurses and physicians of the intensive care units of a Portuguese hospital center (N=275). The inclusion criteria were, to be a nurse or a physician, to provide care in a intensive care unit of the identified hospital center (cirurgical, cardiothoracic, coronary, medical or trauma). On the other hand, the exclusion criteria were, be any other health professional, providing care in settings other than intensive care settings, absence of informed consent, belonging to the invited group of experts, participation in the instrument design pre-test.

Participants were invited via institutional email and data was collected through the access of on-line platforms.

The experimental group was asked to use the game. Two weeks were defined as the time to use the game. The use of the game can be seen by the coded digital record on its digital platform. The control group neither used nor had access to the game. Afterwards both groups performed the ALS knowledge assessment test. It is a test with 20 multiple choice questions each scored as right (0.5 points) or wrong (0 points).

The sample was stratified in order to eliminate "professional group" variable. This was a protocol update at made at 10th of March

ELIGIBILITY:
Inclusion Criteria:

* to be a nurse or a physician,
* to provide care in a intensive care unit of the identified hospital center (cirurgical, cardiothoracic, coronary, medical or trauma)

Exclusion Criteria:

* be any other health professional
* providing care in settings other than intensive care settings
* absence of informed consent
* belonging to the invited group of experts
* participation in the instrument design pre-test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
The score at the advanced life support knowledge assessment test | 3 weeks
  The minimun score at the scale is 0 and the maximum is 100, were 100 means the best result.
  It was applied through an online application, facilitating the participation of the guests and providing the automatic transcription of the results. The platform registration was carried out in a coded manner, thus ensuring the anonymity of the participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Chvng, Vila Nova de Gaia, Portugal